CLINICAL TRIAL: NCT07072598
Title: Comparing Efficiency and Stone-Free Rates After Mini-Percutaneous Nephrolithotomy and Flexible Ureteroscopy With Suction Access Sheaths
Brief Title: Comparing Efficiency and Stone-Free Rates Mini PCNL vs Flex URS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: KARL STORZ Endoscopy-America, Inc. (Industry)
Responsible Party: Principal Investigator, Amy Krambeck, Director of the Endourology/Stone Division, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00222993
Record Dates: First submitted 2025-06-24; First posted 2025-07-18 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-07

CONDITIONS: Kidney Stones; Nephrolithiasis; Urolithiasis
Keywords: kidney stone; Ureteroscopy; Mini-PCNL; ClearPETRA; kidney stone interventional treatment; kidney stone 1cm-3cm
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis; Urolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Ureteroscopy (Active Comparator): Patients randomized to this arm will have their stones treated using the method of Ureteroscopy in a standardized fashion. A second 0.035in sensor guidewire will then be advanced up to the renal pelvis with placement confirmed by fluoroscopy. Placement of a 12/14Fr ClearPETRA ureteral access sheath will be attempted. If this is unsuccessful, a 11/13Fr ClearPETRA ureteral access sheath will be advanced over the wire. If this is unsuccessful, a 5Fr open ended ureteral catheter will be placed and procedure will be converted to a miniPCNL. Lithotripsy will be performed with the MOSES 2.0 high power Holmium laser with settings of 0.3J and 120Hz or 2J and 20Hz depending on stone location and appearance. Stones will be extracted with the suction access sheath. A ureteral stent will be placed at the conclusion of the procedure.
  Interventions: Device: ClearPETRA suction access sheath
- Mini-PCNL (Active Comparator): Will be performed by first starting with supine flexible cystoscopy to cannulate the ureteral orifice with a 5Fr open ended ureteral catheter. The patient will then be repositioned prone with 1-2 bumps placed transversely across the chest. Contrast will be instilled into the ureteral catheter and renal access will be obtained fluoroscopically with the triangulation technique. Once access is obtained, the tract will be dilated to 20Fr and a 18/20Fr ClearPETRA renal access sheath will be inserted to assess the collecting system. If there is concern that the 20Fr access is not sufficient to clear the stone, the tract will be upsized to 24 or 30Fr. The stones will be evacuated with the Trilogy Lithotripter and/or laser, suction and/or basket extraction. A ureteral stent will be placed at the conclusion of the procedure.
  Interventions: Device: ClearPETRA suction access sheath

INTERVENTIONS:
Device: ClearPETRA suction access sheath — Ureteroscopy utilizing the ClearPETRA suction access sheath.
  Arms: Ureteroscopy
Device: ClearPETRA suction access sheath — Mini-PCNL utilizing the ClearPETRA suction access sheath
  Arms: Mini-PCNL

SUMMARY:
The objective of the study is to compare the stone free rates with ureteroscopy utilizing the ClearPETRA suction ureteral access sheath, and mini-PCNL; both procedures and ClearPETRA sheaths are standard of care and are used regularly for stone treatment. Our primary objective is to assess the complete stone free rate with both procedures.

DETAILED DESCRIPTION:
With the advent of mini-PCNLs, some endourologists have been utilizing the technique to treat renal calculi up to 3cm in size with better stone free rates and similar comorbidity compared to ureteroscopy. These procedures require percutaneous renal access, and it is associated with greater length of stay and fluoroscopy time.

The ClearPETRA ureteral access sheath has shown great promise with improving stone free rates, decreasing intra-renal pressure and delivering some of the benefits of mini-PCNL without the added risk associated with obtaining percutaneous renal access.

The ClearPETRA flexible suction ureteral access sheath anecdotally improves efficiency and allows endourologists to better clear stone debris when compared to traditional ureteral access sheaths. We have yet to see a comparison between suction ureteral access sheaths and mini-PCNL with the suction renal access sheath.

Study Hypothesis: Compared to traditional access sheaths, using ClearPETRA access sheaths will result in an improvement in stone free rates with both modalities, with lower complications. Using ClearPETRA access sheaths in both modalities compared to traditional access sheaths should result in less of a difference in stone free rates between the ureteroscopy group and the mini-PCNL group.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Have a CT scan showing renal stones 1-3cm in length
* Patients who will be able to read, understand, and complete patient questionnaires

Exclusion Criteria:

* Pregnant individuals
* Those with anomalous renal anatomy
* Patients with a urinary diversion (ex: Ileal conduit, reservoir, bladder substitute, etc.)
* Any condition rendering patient medically unfit to undergo either procedure (Bleeding diasthesis)
* Patients who lack decisional capacity
* Patients who are non-english speakers*

  * Non-recruitment of non-english speakers is due to the study being a small pilot study that is used to assess the stone free rate for patients treated with a ureteroscopy or mini-PCNL using ClearPETRA suction access sheaths in a small portion of our patient population seeking treatment for stones. The team also does not possess the bandwidth or personnel to consent patients who are non-English speaking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Stone free rate | 4 weeks post-procedure
  Stone free rate (no residual stone) on post-procedure CT

SECONDARY OUTCOMES:
Surgery time | Procedure day (1 day)
  Surgery time (minutes)
Complication rate | Procedure day (1 day)
  Complication rate (Clavien-Dindo) (%)
Unplanned hospital visits | 90 days postoperatively
  Unplanned hospital visits (ED/clinic)
Need for additional procedure | 90 days postoperatively
  Need for additional procedure (within 90 days postoperatively)
Length of stay | Perioperatively (starting at Baseline/Procedure Date)
  Length of stay hospital stay (if admitted post-procedure, or readmitted)
Inability to access ureter | Procedure day (1 day)
  Intra-operative complications including inability to access the ureter ureteroscopically or need to upsize the renal access sheath with the percutaneous approach.
Need to upsize from 18Fr Sheath | Procedure day (1 day)
  Need to upsize from 18Fr (PCNL group)
Occurrence of post-procedure sepsis | Perioperatively (starting at Baseline/Procedure Date)
  Post-op sepsis
Hospital / patient costs (in total for procedure and any necessary postoperative hospital admissions or procedures related to the initial procedure). | Perioperatively (starting at Baseline/Procedure Date)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States